CLINICAL TRIAL: NCT04823481
Title: Acute Anterior or Posterior Cerebral Artery Occlusion Recanalization Therapy and Relationships With Clinical Outcome (ACAPULCO)
Acronym: ACAPULCO
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: CE_20210126_8_PSS
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Ischemic Stroke; Thrombi
MeSH Terms: conditions — Ischemic Stroke; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nearly 3% of patients with ischaemic stroke (IS) have an isolated occlusion of the anterior or posterior cerebral artery in the acute phase of the disease. In those patients, intravenous thrombolysis (IT) is indicated for 4.5 hours after symptoms onset. Due to a lack of data, mechanical thrombectomy (MT) is not considered as a gold standard to treat IS alone or in addition with IT. Therefore, observational studies are needed to understand the clinical evolution of patients with IS treated with IT and/or MT. The ACAPULCO retrospective observational study aims to highlight potential benefits of MT in those patients to improve their management and to propose targeted therapies in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and < 96
* Clinical signs consistent with acute ischemic stroke
* Patients who presented within 6 hours of stroke symptoms onset
* Isolated occlusion of the anterior or the posterior artery

Exclusion Criteria:

* Administration of recanalization treatment before hospital admission

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects having clinical signs and imaging criteria consistent with acute ischemic stroke who presented within 6 hours of stroke symptoms onset with isolated occlusion of the anterior or the posterior artery.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Clinico-radiological evolution of IS patients with isolated occlusion of the anterior or posterior cerebral artery. | 90 days
  Good Neurological Condition Good neurological outcome (GNO) at 3 months will defined using the modified Rankin Scale (mRS). A normal/near normal outcome after procedure is associated with a mRS Scale score = 0-1 and severe disability/death is associated with a mRS Scale score = 5-6

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Seners, MD,PhD, Principal Investigator — Hôpital Fondation Adolphe de Rothschild
Locations (1):
- Hôpital Fondation Adolphe de Rothschild, Paris, Île-de-France Region, France